CLINICAL TRIAL: NCT07210918
Title: Serum Trace Element Profiles in Women With Endometriosis, Ovarian and Endometrial Cancer: An ICP-MS-Based Comparative Study
Brief Title: Serum Trace Element Levels in Some Gynecological Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Dilara Ulger Ozbek, Dr., Cumhuriyet University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Cütam Dilara
Record Dates: First submitted 2025-09-30; First posted 2025-10-07 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Endometriosis; Endometrial Cancer; Over Cancer; Healthy Control
Keywords: trace elements; endometriosis; endometrial cancer; overian cancer
MeSH Terms: conditions — Endometriosis; Endometrial Neoplasms

STUDY DESIGN:
Intervention Model Description: We have four groups in the study. Blood will be drawn from each group only once. No other interventions will be performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group (Experimental): Consists of healthy individuals
  Interventions: Diagnostic Test: Blood Product
- Endometriosis group (Experimental): Consists of individuals diagnosed with endometriosis
  Interventions: Diagnostic Test: Blood Product
- Overian cancer group (Experimental): Consists of individuals diagnosed with ovarian cancer
  Interventions: Diagnostic Test: Blood Product
- Endometrial cancer (Experimental): Consists of individuals diagnosed with endometrial cancer
  Interventions: Diagnostic Test: Blood Product

INTERVENTIONS:
Diagnostic Test: Blood Product — 5 mL of blood was collected from the right arms of all individuals in 4 different groups. Their serum was obtained.

SUMMARY:
The aim of this clinical study is to measure the levels of various trace elements in the blood serum of women with various gynecological diseases and to compare them with healthy controls. The main questions it aims to answer are:

* Do trace element levels increase or decrease in endometriosis?
* Do trace element levels increase or decrease in ovarian cancer patients?
* Do trace element levels increase or decrease in endometrial cancer patients?

Participants:

Each member of the study group will visit the clinic only once and donate 5 ml of blood.

DETAILED DESCRIPTION:
However, the serum trace elements profiles of individuals with endometriosis, ovarian cancer (OC), and endometrial cancer (EC) are not fully known. The purpose of this study is to examine the levels of trace element profiles in the blood serum of healthy people and individuals with gynecological disorders.

The study group comprised of 40 women divided into four groups (n=10 each); endometriosis, endometrial cancer and ovarian cancer, and control group who were obstetrically and demographically similar. Inductively coupled plasma-mass spectrometry (ICP-MS) was used to assess serum trace element levels of lead, beryllium, vanadium, chromium, manganese, iron, cobalt, nickel, arsenic, selenium, molybdenum, cadmium, antimony, and phosphorus

ELIGIBILITY:
Inclusion Criteria:

* Not having received chemotherapy, radiotherapy or immunotherapy in the last three months
* For the endometriosis group: histopathologically or laparoscopically confirmed endometriosis
* For the ovarian cancer group: histopathologically confirmed epithelial ovarian cancer
* For the endometrial cancer group: histopathologically confirmed endometrial adenocarcinoma
* For the control group: healthy individuals who underwent surgery for benign gynecological causes (e.g., myoma, benign cyst) and who were not diagnosed with malignancy/endometriosis

Exclusion Criteria:

* Chronic systemic diseases (e.g., chronic renal failure, liver disease, severe cardiac disease)
* Diseases that may affect metabolism or trace element levels (e.g., Wilson's disease, hemochromatosis)
* Use of dietary supplements containing minerals or trace elements within the past 6 months
* Environmental or occupational heavy metal exposure (e.g., mining, metallurgy, battery industry workers)
* Pregnancy or breastfeeding
* History of acute infection or inflammatory disease
* History of recurrent surgery or advanced metastatic cancer (as this may alter serum parameters)
* Psychiatric or cognitive disorders that preclude participation in the study

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Since this study is about gynecological diseases, female participants must be selected.
Enrollment: 40 (Actual)
Dates: Start 2025-04-24 (Actual); Primary Completion 2025-09-29 (Actual); Study Completion 2025-09-29 (Actual)

PRIMARY OUTCOMES:
Serum beryllium (Be) measurment | 3 months
  Measured beryllium (Be) levels in the serum samples of study group by ICP-MS baseline.
Serum phosphorus (P) measurment | 3 months
  Phosphorus levels (ppb) in the serum samples of study group by ICP-MS baseline.
Serum vanadium (V) mesurment | 3 months
  Measured vanadium (V) levels (ppb) in the serum samples of study group by ICP-MS baseline.
Serum chromium (Cr) measurment | 3 months
  Measured chromium (Cr) levels in the serum samples of study group by ICP-MS baseline.
Serum manganese (Mn) measurment | 3 months
  Measured manganese (Mn) levels in the serum samples of study group by ICP-MS baseline.
Serum iron (Fe) measurment | 3 months
  Measured iron (Fe) levels in the serum samples of study group by ICP-MS baseline.
Serum cobalt (Co) measurment | 3 months
  Measured cobalt (Co) levels in the serum samples of study group by ICP-MS baseline.
Serum nickel (Ni) measurment | 3 months
  Measured nickel (Ni) levels in the serum samples of study group by ICP-MS baseline.
Serum arsenic (As) measurment | 3 months
  Measured arsenic (As) levels in the serum samples of study group by ICP-MS baseline.
Serum selenium (Se) measurment | 3 months
  Measured selenium (Se) levels in the serum samples of study group by ICP-MS baseline.
Serum molybdenum (Mo) measurment | 3 months
  Measured molybdenum (Mo) levels in the serum samples of study group by ICP-MS baseline.
Serum cadmium (Cd) measurment | 3 months
  Measured cadmium (Cd) levels in the serum samples of study group by ICP-MS baseline.
Serum antimony (Sb) measurment | 3 months
  Measured antimony (Sb) levels in the serum samples of study group by ICP-MS baseline.
Serum lead (Pb) measurment | 3 months
  Measured lead (Pb) levels in the serum samples of study group by ICP-MS baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- sivas Cumhuriyet University, Sivas, Centre, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No